CLINICAL TRIAL: NCT03077789
Title: Prospective Study of the Diagnostic and Therapeutic Management of Congenital Glaucoma in France
Acronym: Conglau
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011_32; 2012-A00929-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Congenital Glaucoma
Keywords: visual acuity; prognosis epidemiology
MeSH Terms: conditions — Hydrophthalmos | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRABECULOTOMY (Experimental)
  Interventions: Procedure: TRABECULOTOMY

INTERVENTIONS:
Procedure: TRABECULOTOMY — Evaluation of the prognosis of different surgery in congenital glaucoma
  Other Names: sclerectomy needling trabeculectomy

SUMMARY:
Evidence of a relationship between age at discovery of congenital glaucoma and visual acuity at 4 years of age.

The delay in diagnosis is a factor of poor visual acuity. Will justify the implementation of information programs with health and education professionals in order to improve the functional prognosis of patients with congenital glaucoma.

DETAILED DESCRIPTION:
Prospective multicentre prospective cohort Enabling the identification and follow-up of an almost exhaustive population of incidents of congenital glaucoma in 23 ophthalmology centers in France Inclusion over 4 years Epidemiological data, all reports of consultation, medical and surgical procedures collected in an E-CRF.

Database for gene research related to congenital glaucoma to provide screening, genetic counseling and personalized care

ELIGIBILITY:
Inclusion Criteria:

* Boys or girls under the age of 4, without antecedent, French or resident in France, Suspected Glaucoma

Exclusion Criteria:

* Antecedent of surgery for glaucoma

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Visual acuity by logarithmic scale of Sander-Zanlonghi | at 4 years of the child
  Evidence of a relationship between age at discovery of congenital glaucoma and visual acuity at 4 years of age

SECONDARY OUTCOMES:
Intraocular pressure | at 4 years of the child
  measure intraocular pressure (Tonopen or Perkins initially, air tonometer or Goldman as soon as possible) for prognosis of congenital glaucoma

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François ROULAND, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (24):
- France (24):
  - Chu Amiens Picardie - Amiens 1, Amiens
  - Chu Amiens Picardie, Amiens
  - Centre Hospitalier Regional D' Angers, Angers
  - CHRU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon Bourgogne, Dijon
  - Chu de Grenoble Alpes, Grenoble
  - CHRU, Hôpital Claude Huriez, Lille
  - Hopital Edouard Herriot - Hcl - Lyon 03, Lyon
  - Aphm Hopital Nord, Marseille
  - CHRU de Montpellier, Montpellier
  - CHU de Montpellier, Montpellier
  - Centre Hospitalier Universitaire, Nantes
  - Chu de Nice Hopital de L'Archet, Nice
  - Fondation de Rothschild - Paris, Paris
  - Hu Necker Enfants Malades Aphp - Paris 15, Paris
  - Hopital Robert Debre Chu Reims, Reims
  - Chru Rennes Site Pontchaillou, Rennes
  - Hopital Charles Nicolle Chu Rouen, Rouen
  - Hopital Civil / Nouvel Hopital Civil - Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHRU de Tours, Tours
  - Chu de Tours, Tours

IPD SHARING:
Plan to Share IPD: No